CLINICAL TRIAL: NCT04476251
Title: A Pilot Study of E7 TCR T Cell Induction Immunotherapy for Stage IIB-IVA Cervical Cancer
Brief Title: E7 TCR T Cell Induction Immunotherapy for Stage IIB-IVA Cervical Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Multiple logistical challenges
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Norberg, D.O., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200116; 20-C-0116
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Uterine Cervical Neoplasms
Keywords: T Cell Receptor; Immunotherapy; Aldesleukin; Cyclophosphamide; Fludarabine
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy (Experimental): E7 TCR T Cell Therapy
  Interventions: Biological: E7 T-Cell Receptor (TCR)

INTERVENTIONS:
Biological: E7 T-Cell Receptor (TCR) — Patients will receive up to 3x10^10 E7 T-Cell Receptor (TCR) T cells (i.e. TCR+ cells).

SUMMARY:
Background:

More than 12,000 cases of cervical cancer are diagnosed in the United States each year. A new therapy has been developed that involves taking white blood cells from a person, genetically modifying the cells in a lab so they recognize cancer, and then giving the cells back to the person. Researchers want to see if this therapy can help people with cervical cancer.

Objective:

To find out if people with Stage IIB-IVA cervical cancer can safely be given E7 T-cell receptor (TCR) T cells before they get standard treatment.

Eligibility:

People age 18 and older who have Stage IIB-IVA cervical cancer

Design:

Participants will be screened under a separate protocol. Tests will include:

* Physical exam
* Medicine review
* Blood tests
* Pregnancy test (if needed)
* Vein assessment
* Tumor sample or biopsy
* Electrocardiogram (to record the hearts electrical activity)
* Imaging scans, x-rays, and/or endoscopy
* Heart and/or lung tests.

Some screening tests will be repeated during the study.

Participants will undergo leukapheresis. For this, blood is removed through a needle in the arm. A machine removes the white blood cells. The rest of the blood is returned through a needle in the other arm. Participants may need to have a large catheter inserted into a vein.

Participants will stay at the hospital for 2-3 weeks. They will get chemotherapy drugs. They will get the E7 TCR T cells as an intravenous infusion. They will get the drug aldesleukin.

Participants will visit the National Institutes of Health (NIH) 3 and 6 weeks after treatment. They will be contacted yearly for 5 years. They will be asked to participate in long-term follow-up for 15 years....

DETAILED DESCRIPTION:
Background:

* Cervical cancer is the third most common cause of death among women with gynecologic cancers in the United States. Worldwide, cervical cancer accounts for nearly 300,000 deaths annually.
* Virtually all cases of cervical cancer result from chronic infection with high-risk human papillomavirus (HPV), the most common type being HPV16.
* The treatment of locally advanced cervical cancer consists of chemoradiation +/- extended field radiation therapy. Participants with International Federation of Gynecology and Obstetrics (FIGO) (revised 2018) stage III-IVA have the worse prognosis with approximately 50% of the participants dying from their disease within 5 years.
* Induction chemotherapy is an active area of study in this type of cancer. The aim of induction therapy is to reduce the risk of disease recurrence and improve overall survival.
* E7 T-cell receptor (TCR) T cells, administered as a single infusion, have demonstrated safety and clinical activity in advanced, treatment-refractory metastatic HPV+ cancers.

Objectives:

-To determine the feasibility of induction E7 TCR T cell therapy for FIGO (2018) stage IIB-IVA, HPV16+ cervical cancer

Eligibility:

* Participants greater than or equal to 18 years old with FIGO (2018) stage IIB-IVA cervical cancer.
* The cancer must be human papillomavirus 16 (HPV16+) and participant must be HLA-A*02:01+.
* Participants must be treatment-naive (i.e., no prior local or systemic treatment, including radiation; prior loop electrosurgical excision procedure (LEEP) procedure or cone biopsy is allowed).

Design:

* This is a single arm, pilot study, testing the feasibility of induction E7 TCR T cell therapy.
* Participants will receive a conditioning regimen of cyclophosphamide and fludarabine, a single infusion of E7 TCR T cells, and systemic aldesleukin.
* Participants will be referred for standard of care definitive therapy (i.e., chemoradiation +/- extended field radiation therapy) within 6 weeks after infusion of E7 TCR T cells.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Participants with histologically or cytologically confirmed carcinoma of the cervix that has not been treated, with clinical staging as follows:

   * Lead-in safety cohort: FIGO (International Federation of Gynecology and Obstetrics) stage IIIC-IVA (2018 International FIGO Staging System)
   * After lead-in safety cohort: FIGO stage IIB-IVA (2018 International FIGO Staging System)
2. Human papillomavirus 16 (HPV16+) tumor and HLA-A*02:01+ Human leukocyte antigen (HLA) type. Note: HLA-A*02 is also acceptable for enrollment but not for treatment.
3. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria or Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) (if not eligible by RECIST 1.1).
4. Age 18 years. Because no dosing or adverse event data are currently available on the use of E7 TCR T cells in participants <18 years of age, children are excluded from this study. Note: This age range is consistent with the age of participants with the disease being studied.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
6. Women of child-bearing potential must have a negative pregnancy test because E7 TCR T cells have unknown potential for teratogenic or abortifacient effects. Women of child- bearing potential are defined as all women who are not post-menopausal or who have not had a hysterectomy. Note: Postmenopausal will be defined in this study as women over the age of 55 who have not had a menstrual period in at least 1 year.
7. The effects of E7 TCR T cells on the developing human fetus are unknown. For this reason and because the chemotherapy agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (e.g., intrauterine device, hormonal or barrier method of birth control; abstinence; tubal ligation or vasectomy) prior to study entry and for four months after treatment. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
8. Seronegative for HIV (human immunodeficiency virus) antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment.
9. Seronegative for hepatitis B antigen and hepatitis C antibody. If hepatitis C antibody test is positive, then the participant must be tested for the presence of antigen by Reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C Virus (HCV) ribonucleic acid (RNA) negative.
10. Must be willing to participate in Gene Therapy Long Term Follow up Protocol (20C0051), which will follow participants for up to 15 years per Food and Drug Administration (FDA) requirements.
11. Participants must have organ and marrow function as defined below:

    * leukocytes >=3,000/mcL
    * absolute neutrophil count >=1,500/mcL
    * platelets >=100,000/mcL
    * hemoglobin >=9.0 g/dL
    * total bilirubin within normal institutional limits except in participants with Gilbert's Syndrome who must have a total bilirubin < 3.0 mg/dL
    * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT) Serum ALT/AST < 2.5X ULN
    * creatinine clearance Calculated creatinine clearance (CrCl) >=50 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)
12. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Previous treatment for invasive cervical cancer including:

   * Chemotherapy or other systemic treatments
   * Radiation therapy
   * Hysterectomy (prior LEEP procedure or cone biopsy is allowed)
2. Participants who are receiving any other investigational agents.
3. History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations at the time of treatment that would limit compliance with study requirements.
5. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR T cells, breastfeeding should be discontinued if the mother is treated with E7 TCR T cells. These potential risks may also apply to other agents used in this study.
6. Participants with any form of systemic immunodeficiency, including acquired deficiency such as HIV or primary immunodeficiency such as Severe Combined Immunodeficiency Disease, are ineligible. The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who have decreased immune competence may be less responsive to the treatment.
7. Participants on immunosuppressive drugs including corticosteroids.
8. Participants with autoimmune diseases such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis, autoimmune pancreatitis, or systemic lupus erythematosus. Hypothyroidism, vitiligo and other minor autoimmune disorders are not exclusionary.
9. Participants with a second invasive malignancy requiring treatment within the last 2 years are not eligible with the following exceptions:

   * Ductal carcinoma in situ (DCIS) of the breast
   * Cutaneous skin cancers requiring only local excision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0116.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy: E7 TCR T Cell Therapy
  E7 TCR: Patients will receive up to 3x10^10 E7 T-Cell Receptor (TCR) T cells (i.e. TCR+ cells).
Period: Overall Study
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Fraction of Participants for Whom E7 T-Cell Receptor (TCR) Induction Therapy is Feasible in Participants With Cervical Cancer
Description: The Fraction of participants for whom E7 T-Cell Receptor (TCR) induction therapy is feasible in participants with cervical cancer
Time Frame: 6 months
Population: This outcome measure was not done due to multiple logistical challenges. One participant was enrolled but not treated.
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Fraction of Participants With Relapse-free Survival at 2 Years and 5 Years Following Definitive Standard of Care Therapy
Description: Fraction of participants with relapse-free survival at 2 years and 5 years estimated from a Kaplan-Meier curve of relapsed free survival following definitive standard of care therapy who achieve a success. Relapsed free survival is defined as the time from date on study to date of relapse of disease.
Time Frame: 2 yrs and 5 yrs
Population: This outcome measure was not done due to multiple logistical challenges. One participant was enrolled but not treated.
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Fraction of Participants With Grade 1-5 Adverse Events
Description: To evaluate the safety of E7 induction therapy, the types and grades of toxicity obtained will be reported. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: 1 year
Population: This outcome measure was not done due to multiple logistical challenges. One participant was enrolled but not treated.
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of E7 T-Cell Receptor (TCR)T Cells Following Completion of Chemoradiation
Description: Percentage of E7 T-Cell Receptor (TCR)T cells following completion of chemoradiation
Time Frame: 1 year
Population: This outcome measure was not done due to multiple logistical challenges. One participant was enrolled but not treated.
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Fraction of Participants Who Achieve an Objective Response (Partial Response + Complete Response) Following E7 T-Cell Receptor (TCR) T Cell Induction Therapy
Description: Fraction of participants who achieve an objective response (Partial Response + Complete Response) following E7 induction therapy will be reported. Response may be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesion; and/or Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST). Complete Metabolic Response is complete resolution of F-fluorodeoxyglucose (FDG) uptake in all lesions, and Partial Metabolic Response is ≥ 30% reduction of the SUL (lean body mass corrected standard uptake value) peak and an absolute drop of 0.8 SULpeak units.
Time Frame: 1 year
Population: This outcome measure was not done due to multiple logistical challenges. One participant was enrolled but not treated.
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 20 days.
Population: This outcome measure was not done due to multiple logistical challenges. One participant was enrolled but not treated.
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 20 days.
Arm/Group | Arm 1/E7 T-Cell Receptor (TCR) T Cell Therapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT04476251/Prot_SAP_000.pdf
  • Informed Consent Form: Screening Consent (2021-01-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT04476251/ICF_001.pdf
  • Informed Consent Form: Affected Patient Consent (2021-01-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT04476251/ICF_002.pdf